CLINICAL TRIAL: NCT02673047
Title: Observational Study of Botulinum Toxin Type A in Patients With Urinary Incontinence Associated With Overactive Bladder
Acronym: BOREAL
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/NS/OAB/006
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Bladder, Overactive; Urinary Bladder, Neurogenic
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder, Neurogenic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Botox®: Patients prescribed botulinum toxin Type A (Botox®) injection for the treatment of urinary incontinence associated with neurogenic detrusor overactivity or overactive bladder as per standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A (Botox®) injection as prescribed as standard of care in clinical practice.
  Other Names: Botox®; onabotulinumtoxinA

SUMMARY:
This study will describe the prescription conditions of botulinum toxin Type A (Botox®) injection for the treatment of urinary incontinence due to neurogenic detrusor overactivity (NDO) or idiopathic overactive bladder (IOAB) as per standard of care in clinical practice in France.

ELIGIBILITY:
Inclusion Criteria:

-Patients who receive a Botox® injection for urinary incontinence.

Exclusion Criteria:

-Patients not residing in France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with Botox® for urinary incontinence associated with NDO or IOAB in clinical practice.
Sampling Method: Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Target Patients Prescribed Botox® in Clinical Practice | Day 1

SECONDARY OUTCOMES:
Treatments Previously Prescribed | Day 1
Number of Sites Injected | Day 1
Total Dose of Botox® Used | Day 1
Types of Anaesthesia and Antibiotic Prophylaxis Used | Day 1
Cytobacteriological Examination of the Urine | Day 1
Total Number of Botox® Cycles in Non-naive Patients (previously received Botox®) | Day 1
Length of Botox® Treatment in Non-naive Patients | Day 1
Time Since Last Botox® Injection in Non-naive Patients | Day 1
Characteristics of Injector Sites (Locations) | Day 1
Characteristics of Injector Physicians | Day 1
Characteristics of Patients | Day 1
Number of Patients by Pathology History | Day 1
Number of Patients by Medical and Surgical History | Day 1
Reduction of Number of Daily Urinary Incontinence Episodes in Non-naive Patients | Day 1
Percentage of Continent Patients in Non-naive Patients | Day 1
Number of Adverse Events during the Visit | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (50):
- France (50):
  - Site D'Aix En Provence, Aix-en-Provence
  - CL Toulouse Lautrec, Albi
  - CHU Angers, Angers
  - CH Angouleme, Angoulême
  - CH Avranches Granville, Avranches
  - CH Bagnols Sur Ceze, Bagnols-sur-Cèze
  - CH Belfort, Belfort
  - CHU Besancon, Besançon
  - CL Saint Augustin, Bordeaux
  - CHU Bordeaux, Bordeaux
  - CH de Cahors, Cahors
  - CH Châlons-en-Champagne, Châlons-en-Champagne
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CH Colmar, Colmar
  - CHU Mondor (APHP), Créteil
  - CH Hopale Ctre Calot/Helio, Cucq
  - CHU Dijon, Dijon
  - CHI E.Durkheim Plateau de La Justice, Épinal
  - CH Raymond Poincare (APHP), Garches
  - CH Renee Sabran Hyeres (HCL), Giens-Hyeres
  - GH de la Rochelle Ré-Aunis, La Rochelle
  - CH Bicêtre (APHP), Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHU Limoges, Limoges
  - CL Mutualiste Porte de L'Orient, Lorient
  - CH de la Conception (APHM), Marseille
  - CH Mont de Marsan, Mont-de-Marsan
  - CL Beau Soleil, Montpellier
  - CHU Montpellier, Montpellier
  - CH Mulhouse, Mulhouse
  - CHU Nimes, Nîmes
  - GH Saint Joseph, Paris
  - CH Tenon (APHP), Paris
  - CH Lyon Sud (HCL), Pierre-Bénite
  - CH de Pontoise, Pointoise Cedex
  - USLD de Lusignan, Poitiers
  - CH Annecy, Pringy
  - SIH Privas La Voulte, Privas
  - Polyclinique Les Bleuets, Reims
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CL de L'Alliance Saint Cyr/Loire, Saint Cyr/Loire
  - CH Saint-Avold, Saint-Avold
  - CL Mutualiste Chirurgicale, Saint-Etienne
  - CH de Saintonge (Saintes), Saintes
  - Hôpital Civil / Nouvel Hôpital Civil, Strasbourg
  - CH Foch, Suresnes
  - Clinique de l'Ormeau Pyrénées, Tarbes
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours